CLINICAL TRIAL: NCT04136379
Title: Comparison of Efficacy and Outcomes for Home and Standard Clinic Monitoring of INR in Patients With Congenital Heart Disease
Brief Title: Comparison of Home and Standard Clinic Monitoring of INR in Patients With CHD
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0081
Record Dates: First submitted 2019-10-07; First posted 2019-10-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Congenital Heart Disease; Congenital Heart Defect; Adult Congenital Heart Disease
Keywords: Warfarin therapy; INR monitoring
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinic monitoring: Patients who attend a warfarin clinic for management of their INR
- Home monitoring: Patients who undertake home monitoring of their INR using a CoaguChek POC device
  Interventions: Diagnostic Test: INR monitoring using a CoaguChek POC device

INTERVENTIONS:
Diagnostic Test: INR monitoring using a CoaguChek POC device — INR monitoring using a CoaguChek POC device
  Groups: Home monitoring

SUMMARY:
Summary: Congenital heart disease (CHD) is the most prevalent form of birth defect with a global rate of 1.35 million newborns born with CHD annually. Patients with CHD have an increased risk of cerebrovascular accident (CVA) compared to age-matched control populations. Anticoagulation with warfarin is the mainstay of antithrombotic treatment in these patients and requires frequent monitoring of the International Normalized Ratio (INR). The CoaguChek monitor is a point of care device that enables patients to self-monitor and manage their INR without the need to attend a warfarin clinic. The aim of this study is to compare the efficacy and outcomes of standard clinic management and home management of INR in patients with CHD. Analysis of time in therapeutic range (TTR), INR variability, major and minor bleeding events, incidence of CVA and other thrombotic events will be undertaken. Original Hypothesis: There will be a difference in the proportion of time that patients spend in their therapeutic range and the amount of adverse events that occur between those who use a CoaguChek monitor and those who use standard clinic monitoring of their INR. The primary outcome will be time in therapeutic range (TTR). Secondary outcomes will be INR variability, minor / major bleeding complications and thromboembolic events.

DETAILED DESCRIPTION:
Aims and Objectives: The aim of this study is to compare the efficacy and outcomes of standard clinic management and home management of INR in patients over 14 years of age with CHD and to determine which method of INR management results in a greater time in therapeutic range, less INR variability and fewer adverse events. This study will have a number of objectives as detailed below.

1. To determine whether patients who home monitor their INR or those who use standard clinic management spend more time in therapeutic range with less INR variability and have fewer adverse events.
2. To survey patient views on the ease of use, practicality and their satisfaction with their current method of INR management.
3. To examine patients overall health related quality of life (HRQoL) using RAND SF-36 survey for participants who are 18+ years and the PedsQL quality of life inventory for participants who are 14-17 years of age, and determine whether there is a difference in HRQoL between the two cohorts.
4. To undertake structured interviews with the participants' General Practitioners (GPs) to examine their views / beliefs about INR home monitoring; and to undertake semi-structured interviews with the ACHD clinical nurse specialists and the clinical research nurse (who is responsible for training patients in the use of home monitoring) to examine their views about INR home monitoring.

Experimental details and design of proposed investigation: This research will be a 1-year prospective cohort study monitoring CHD patients who are on warfarin. Recruitment of patients will be from the ACHD clinics in the Royal Victoria Hospital (RVH), Belfast. There are approximately 4,000 patients with CHD who attend these clinics from the age of 14 years onwards, with a proportion of these patients on warfarin therapy. Patients on warfarin will be identified by Jan Gordon (ACHD clinical nurse specialist) or Deirdre Lovell (clinical research nurse). Suitable patients who attend one of the ACHD clinics during the 6 month recruitment period will be sent a participant information leaflet at the same time as they are sent their clinic appointment letter (which is sent out two weeks prior to their appointment). Eligible participants can also be recruited from other clinics in RVH. The participant information sheet will inform them about the study and contain contact information for the PhD student, Rachel Savage, who can provide more information and explain the study further. Interested patients will have two weeks to consider their participation prior to their clinic appointment. The PhD student will attend the ACHD clinics up to three times per week for six months to explain the study and recruit patients. Dr Lockhart (Adult CHD Consultant) and Jan Gordon will support this recruitment process. Patients who agree to participate in the study will be screened for inclusion / exclusion criteria as detailed below, and if eligible be asked to provide informed consent. Inpatients who meet the eligibility criteria will be identified by a clinical member of the research team, and provided with the participant information sheet. Those who are interested in participating in the study will notify one of the clinical member of the research team, in which case the PhD student will be informed, and will attend the RVH to gain informed consent allowing at least one week to consider their participation.

There is currently a home monitoring programme at the RVH which is run by a nurse specialist who trains patients how to use their CoaguChek monitor and how to self manage their warfarin dose, following the RVH protocols regarding frequency of testing and dose adjustment. After a 4 month training period, long term follow up of these patients is undertaken by their GP. There is a proportion of ACHD patients who currently home monitor using the RVH protocols. In the event of any issues with home monitoring, patients can contact their GP or one of the ACHD clinical nurse specialists for advice. The patients who currently home monitor will have chosen to home monitor and will either have purchased the CoaguChek monitor themselves, or will have received a monitor which has been funded by Children's Heartbeat Trust, who provide funding for 15 new monitors for ACHD patients per year.

Data Collection: Patients in both cohorts will be asked to submit an electronic INR record, which includes their INR level, warfarin dose, acute illnesses, changes in medications and any warfarin-related adverse events e.g. minor / major bleeding and thromboembolic events, as per normal practice. Acute illnesses and changes in medications are potential covariates and will be included in covariate analysis. Additionally alcohol intake is a potential covariate, which will be recorded at recruitment. An email and/or text message will be sent to all participants at the end of each month to remind them to submit their INR record electronically to Rachel Savage. Participants in the home monitoring cohort will be invited to attend the RVH at 6 months and at the end of the 12 months to have their INR data downloaded from their CoaguChek monitor. Data for the standard clinic monitoring cohort will also be obtained at 6 months and again at 12 months, from the participants' electronic health record (ECR), by either the clinical research nurse or one of the ACHD clinical nurse specialists within the Belfast Health and Social Care Trust. In cases of suspected CVA, the CT/MRI will be reviewed by a Consultant Radiologist as per normal clinical practice.

At the end of the twelve month follow up period all participants will be asked to complete a patient satisfaction questionnaire, which will evaluate the ease of use, practicality and their satisfaction with the method of INR management they use. Questions will include, but are not limited to the following: indication for warfarin therapy, INR target range, duration of warfarin therapy, history of blood clots/stroke/TIA, history of INR levels <1.5 or >8 and how often their INR is checked. A link to the patient questionnaire will be sent electronically to all participants at the end of the study.

Participants who are 18+ years will be asked to complete a health related quality of life (HRQoL) survey RAND SF-36, to determine whether home management of INR affects quality of life. A link to the HRQoL survey will be sent electronically to all participants who are 18+ years at the end of the 12 month follow up period. For participants who are 14-17 years, the PedsQL inventory will be used, which is a validated, disease-specific questionnaire for use by paediatric patients. At the end of the twelve month follow up period, an electronic link to the PedsQL inventory will be sent to participants who are 14-17 years.

Each participant's General Practitioner (GP) will be invited to take part in structured interviews to examine their views / beliefs regarding INR home monitoring. If there is a GP in the practice who specializes in warfarin monitoring, this GP will also be invited to take part in structured interviews. The aim of the interviews is to determine GP's views on INR monitoring and to examine whether GP preferences influence the method of INR monitoring that patients choose. The participant information sheet and consent form will be sent to each GP along with the letter informing them that their patient is participating in the cohort study. If a GP consents to participate in a structured interview, the PhD student will arrange a suitable time and/or venue to conduct the interviews either face to face or via telephone. All interviews will be audio recorded.

The ACHD clinical nurse specialists and the clinical research nurse responsible for training patients how to home monitor will be invited to participate in semi-structured interviews, which will take place face to face. The aim of these interviews is to determine the views and preferences of clinical nurses on INR monitoring and to examine whether these preferences influence the method of INR monitoring that patients choose. A participant information sheet will be given to the nurses during the 6 month recruitment period of the ACHD participants. All interviews will be audio recorded.

Data Analysis: Patient reported INR results will be cross-referenced with INR results downloaded from the CoaguChek monitor (home monitoring cohort) or the participants' electronic health record (clinic monitoring cohort), and data will be input into SPSS for analysis. To determine if there are differences in patient characteristics between cohorts, categories such as gender, age, indication for warfarin therapy as well as levels of education, work and income will be compared. Normality will be tested using the Shapiro-Wilk test. Categorical variables such as number of adverse events will be displayed as frequency/percentages and statistical significance will be determined using chi-square. Continuous variables such as time in therapeutic range will be displayed as mean ± SD and statistical significance will be determined using t-test. Covariates such as alcohol intake, acute illnesses and changes in medications will be analyzed using ANCOVA.

ELIGIBILITY:
Home monitoring cohort

Inclusion Criteria:

* 14+ years old
* Adult Congenital Heart Disease (ACHD)
* attend a clinic in the RVH
* Able to understand, speak, read and write in English
* Patients who currently home manage their INR using a CoaguChek system and are able to submit information electronically

Exclusion Criteria:

* Patients using a CoaguChek S monitor, as this is an older monitor which uses a different mechanism to measure INR compared with the newer models
* Patients who have been using a CoaguChek <6 months.
* Patients who are cyanotic will be excluded if their haematocrit is >55
* Patients who are pregnant will be excluded as warfarin is not prescribed during the first and third trimesters of pregnancy.

Clinic monitoring cohort

Inclusion Criteria:

* 14+ years, have ACHD
* Attend a clinic in the RVH
* Able to understand, speak, read and write in English
* INR managed by a warfarin clinic
* Able to submit information electronically

Exclusion Criteria

* Patients who have been on warfarin <6 months.
* Patients who are pregnant will be excluded as warfarin is not prescribed during the first and third trimesters of pregnancy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attend an ACHD clinic in the Royal Victoria Hospital, Belfast
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Time in therapeutic range (TTR) | 12 months
  The time the patient remains within their therapeutic INR range

SECONDARY OUTCOMES:
INR variability | 12 months
  Absolute difference in consecutive INR results
Number of Adverse events | 12 months
  Number of thromboembolic or haemorrhage events
Patient satisfaction | 12 months
  How satisfied patients are with their current method of INR management examined using a patient satisfaction questionnaire
Health related quality of life (HRQoL): Health related quality of life scores | 12 months
  Health related quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Hughes, PhD, Principal Investigator — Ulster University
Locations (1):
- Royal Victoria Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No